CLINICAL TRIAL: NCT02190773
Title: Effect of Surgical Periodontal Therapy on the RANKL/OPG System : Do we Need Osteo-immune Modulation Targeting RANKL?
Brief Title: Effect of Surgical Therapy on RANKL/OPG (Osteoprotegerin) System
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ezel Berker, Ezel Berker, Hacettepe University
Other Study IDs: RANKL
Record Dates: First submitted 2014-07-08; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Periodontitis; Aggressive Periodontitis; RANKL/OPG Ratio; Gingival Crevicular Fluid
Keywords: Chronic Periodontitis, Aggressive Periodontitis, RANKL/OPG ratio, Gingival crevicular fluid
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Gingival Crevicular fluid (GCF) is collected at baseline and 3 months after the surgical treatment.

GROUPS / COHORTS (3):
- Chronic periodontitis: Surgical periodontal treatment and GCF collection 3 months after treatment
- Agressive periodontitis: Surgical periodontal treatment and GCF collection 3 months after treatment.
- Control group: Periodontally healthy individuals

SUMMARY:
In the present clinical study including chronic, aggressive periodontitis and healthy individuals, the investigators aimed to determine the RANKL, osteoprotegrin (OPG), Interleukin-1 (IL-1β), IL-10, IL-1β levels in gingival crevicular fluid(GCF) before and after surgical periodontal treatment and search out the relationship of clinical parameters with these cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

* Chronic periodontitis having at least 5mm or more probing depth and aggressive periodontitis patients.

Exclusion Criteria:

* Any known systemic disorder, used antibiotics and/or anti-inflammatory medications, had periodontal treatment in the last 3 months and all of them were non smokers. Subjects who were lactating and pregnant were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individulas that applied to periodontology clinic in faculty of dentistry, Hacettepe University.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
RANKL (pmol) level in GCF | Baseline-3 months
  Changes in RANKL levels 3 months after surgical periodontal treatment in Chronic and Aggressive periodontitis determined by ELISA
OPG level (pg) in GCF | Baseline-3 months
  Changes in OPG levels 3 months after surgical periodontal treatment in Chronic and Aggressive periodontitis determined by ELISA
RANKL/OPG ratio | Baseline - 3months
  RANKL/OPG ratio changes 3 months after surgical periodontal treatment in Chronic and Aggressive periodontitis

SECONDARY OUTCOMES:
IL-1β (pg) levels in GCF | Baseline, 3 months after treatment
  Changes in IL-1β levels (determined by ELISA) 3 months after surgical periodontal treatment in Chronic and Aggressive Periodontitis groups
Il-10 (pg) levels in GCF | Baseline-3 months
  Changes in IL-10 levels (determined by ELISA) 3 months after surgical periodontal treatment in Chronic and Aggressive periodontitis

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)